CLINICAL TRIAL: NCT02286414
Title: Benefit/Risk in Real Life of New Oral Anticoagulants and Vitamin K Antagonists in the Treatment of Non Valvular Atrial Fibrillation in Patients Aged 80 Years and Over, Living at Home or in Nursing Home. A Prospective Cohort Study
Brief Title: Benefit/Risk in Real Life of New Oral Anticoagulants and Vitamin K Antagonists in Patients Aged 80 Years and Over
Acronym: PRESAGE-ACO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM13472
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation
Keywords: oral anticoagulants; Geriatrics; General Practitioner; Safety; Misuse
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; apixaban; fluindione; Acenocoumarol; acarboxyprothrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposed group: Patients recieving direct oral anticoagulants (DOA)
  Interventions: Drug: Direct oral antocoagulant: dabigatran, rivaroxaban, apixaban
- Non-exposed group: Patients recieving vitamine K antagonists (VKA)
  Interventions: Drug: Vitamin K antagonist: warfarin, fluindione, acenocoumarol

INTERVENTIONS:
Drug: Direct oral antocoagulant: dabigatran, rivaroxaban, apixaban — Exposure to direct oral antocoagulants : dabigatran, rivaroxaban, apixaban
  Other Names: Direct oral antocoagulant
  Groups: Exposed group
Drug: Vitamin K antagonist: warfarin, fluindione, acenocoumarol — Exposure to vitamin K antagonist
  Other Names: Vitamin K antagonist
  Groups: Non-exposed group

SUMMARY:
The aim of the study is to compare, in real life, the risk benefit (including both major bleeding and thrombotic events (TE) and death from any cause) associated with direct oral anticoagulants (DOA) and with anti vitamin K (VKA) in older adults (≥ 80 years) suffering from non valvular atrial fibrillation and living in community or nursing home settings.

An observational multicenter prospective inception cohort will be conducted within the PRESAGE-Network, an ongoing active network on drug safety in older adults in France involving a sample of general practitioners (GPs) and pharmacists, for an active surveillance of drug safety in older adults. GPs and pharmacists will prospectively include all octo+ patients they care for, newly treated with an oral anticoagulant (VKA or DOA) for nv AF and will follow them during 2 years at least.

DETAILED DESCRIPTION:
* Context: Oral anticoagulation is recommended for prevention of stroke and thrombo-embolic events in people aged 80 years and over (octo+) suffering from non vavular atrial fibrillation (nv AF) and without contraindication to anticoagulant therapy. Two drug classes are available to achieve this oral anticoagulation: the vitaminK antagonists (VKA, warfarin, fluindione and acenocoumarol) or the direct oral anticoagulants (DOA, dabigatran, rivaroxaban and apixaban). The data of evidence-based and post-marketing literature on the benefit/risk ratio of DOA comparatively to VKA are limited, conflicting, potentially biased and finally inconclusive in this population. Nevertheless, octo+ are the age bracket the most at risk for nv AF and the population with the highest risk of both anticoagulant-related major bleedings and AF-related thrombotic (TE) events.
* Objectives: The aim of the study is to assess and compare the real benefits and harms of the two therapeutic strategies available in routine practice, for the anticoagulation in octo+ suffering from nvAF. The main objective is to estimate and compare a composite event including major bleeding, TE events and death from any cause of DOA and VKA in octo+ suffering from nv AF and living in community or nursing home settings. The secondary objectives are, in this population: to estimate and compare the composite event of each DOA (dabigatran, rivaroxaban, and apixaban) with the composite event of VKA, to estimate and compare the rate of occurrence of each component of the composite event in patients exposed to DOA as compared to patients exposed to VKA, to identify factors associated with the occurrence of major bleeding events and TE events in patients exposed to oral anticoagulants (OAC), to describe others adverse drug reactions (ADRs) (not serious bleeding and TE events; other serious or not serious ADRs) and to provide related rates in users of VKA and DOA as well as individual DOA, to describe the utilization patterns of oral anticoagulants.
* Design: An observational multicenter prospective inception cohort will be conducted within the PRESAGE-Network, an ongoing active network on drug safety in older adults in France involving a sample of general practitioners (GPs) and pharmacists, for an active surveillance of drug safety in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 80 years and over
* Newly treated with oral anticoagulants (DOA or VKA) for nv AF (whatever its type) or for flutter
* Living in community or in nursing home
* And consulting a general practionner (GP) and/or a pharmacist participating to the Presage network

Exclusion Criteria:

* Opposition of the patient to the collection of his personal data
* Follow-up deemed impossible

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Consecutive patients aged 80 years or more, newly treated with oral anticoagulants for nv AF or for flutter, living in community or in nursing home
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Composite of major bleeding events or thromboembolic events or death from any cause | 2 years at least
  Major bleeding is defined as a bleeding resulting in death, requiring hospital admission, resulting in persistent or significant disability/incapacity, or being life threatening, according to the WHO definition of seriousness of Adverse Drug Reactions (ADRs). Thromboembolic events (TE) include: Ischemic stroke, systemic or pulmonary embolism.

SECONDARY OUTCOMES:
Major bleeding eventThromboembolic event | 2 years at least
  Bleeding resulting in death, requiring hospital admission, resulting in persistent or significant disability/incapacity, or being life threatening, according to the WHO definition of seriousness of Adverse Drug Reactions (ADRs)
Thromboembolic event | 2 years at least
  Ischemic stroke, systemic or pulmonary embolism
All adverse events | 2 years at least
  All adverse events
Risk factors of TE events or major bleeding events | 2 years at least
  Risk factors of TE events or major bleeding events
Patterns of use of oral anticoagulants | 2 years at least
  Pattern of use will be described by: characteristics of the treated population (age, comorbidities), drug indication, dose and regimen, time on treatment, reason of discontinuation where applicable, concomitant drugs

CONTACTS AND LOCATIONS:
Overall Officials: Florence Tubach, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris, Paris, France